| <b>₹</b> Pfizer C | CLINICAL AND MEDICAL CONTROLLED DOCUMENT (CMCD) REQUIRED FORM/TEMPLATE | | |
|---|---|---|---|
| Identifier | Version | Title | Effective Date |
| CT24-WI-GL02- | 2.0 | SUMMARY OF CHANGES IN | 01-Jun-2022 |
| RF07 | | AMENDED NON-INTERVENTIONAL | |
| | | STUDY PROTOCOL | |

Protocol #: C4221028

OCEANMIST - Comparative effectiveness of different targeted therapies for BRAF-mutated unresectable/metastatic melanoma in the United States



## SUMMARY OF CHANGES IN AMENDED NON-INTERVENTIONAL STUDY PROTOCOL

This amended protocol describes a revised approach for assessment of comparative effectiveness of encorafenib plus binimetinib relative to other targeted therapies for BRAF-mutated unresectable/metastatic melanoma. Analyses conducted based on the originally submitted protocol for study C4221028 were limited to descriptive and unadjusted analyses of real-world data from Flatiron Health, as the sample size of the identified encorafenib plus binimetinib study cohort was judged to be too small for conduct of adjusted comparative effectiveness analyses. Based on the findings of a recently completed study (*Protocol #C4221035: Overall survival (OS) in patients with metastatic BRAFV600-mutant melanoma treated with encorafenib plus binimetinib in the COLUMBUS trial versus in real-world practice data)*, which showed consistent OS outcomes between the COLUMBUS trial Flatiron Health after accounting for differences in patient profiles, in this amended protocol, to enrich the sample size for the encorafenib plus binimetinib combination cohort, data will be pooled across Flatiron and COLUMBUS, and compared versus real-world data for other targeted therapies as described further below.

Key elements of the revised approach are summarized below:

- 1. Pooling of data for encorafenib + binimetinib patients across the phase 3 COLUMBUS trial and the Flatiron Health real-world database: The pooling of data for encorafenib + binimetinib patients across these two sources is justified by the results of study C4221035, which showed, that after harmonizing key patient selection criteria, adjusting for differences in baseline characteristics, and imputing missing data on baseline characteristics, OS for metastatic BRAFV600-mutant melanoma patients was similar across the COLUMBUS trial and real-world practice data from the Flatiron Health database (HR = 1.03, 95% CI: 0.53, 1.54; p=0.90). Given this empirical consistency in OS outcomes, pooling patients across these settings can be justified and allows for a larger sample size for assessment of comparative effectiveness of encorafenib + binimetinib versus other targeted therapies.
- 2. Application of key patient selection criteria consistent with the COLUMBUS trial for all treatment groups: To ensure included patient populations are comparable across settings, key patient selection criteria applied from the COLUMBUS trial will also be applied to all treatment groups drawn from the Flatiron real-world database. These include the following: age ≥18 years at initiation of targeted therapy, metastatic BRAF V600E/K mutated melanoma without central nervous system metastases, untreated or with prior first-line immunotherapy, and ECOG performance status of 0 or 1.
- Imputation of missing data on baseline characteristics: To allow for more
  comprehensive adjustment for confounding due to differences in baseline characteristics
  between treatment groups, multiple imputation will be conducted to account for missing
  data in baseline characteristics.



The approach outlined here largely follows the approach described in *Protocol #C4221035*, with minor updates to the selection criteria, adjustment factors and statistical methods following discussions with a clinical expert in melanoma and further review of the clinical trial and real-world data.

# Classification of Change as Substantial and Non-Substantial and Rationale

This is a Substantial Protocol Amendment for the reasons described above.



## NON-INTERVENTIONAL (NI) STUDY PROTOCOL

## Study information

| Title | OCEANMIST - Comparative effectiveness of different targeted therapies for BRAF-mutated unresectable/metastatic melanoma in the United States |
|---|---|
| Protocol number | C4221028 |
| Protocol version identifier | 2.0 |
| Date | 19 JUL 2023 |
| Active substance | Encorafenib plus Binimetinib |
| Medicinal product | Braftovi ® plus Mektovi® |
| Research question and objectives | The study objective is to describe and compare OS in patients with metastatic BRAFV600-mutant melanoma treated with encorafenib plus binimetinib (ENCO+BINI) versus other targeted therapies. |
| Author(s) | PPD PharmD, MS PPD ScD PPD Analysis Group, Inc. PPD PhD PPD , Analysis Group, Inc. |
| | PPD , ScD PPD , Analysis Group, Inc. PPD PhD PPD , Analysis Group, Inc. PPD , Analysis Group, Inc. |

This document contains confidential information belonging to Pfizer. Except as otherwise agreed to in writing, by accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others (except where required by applicable law) or use it for unauthorized purposes. In the event of any actual or suspected breach of this obligation, Pfizer must be promptly notified.



| 1. TABLE OF CONTENTS | |
|------------------------------------------------------------------------|----|
| 1. TABLE OF CONTENTS | 5 |
| 2. LIST OF ABBREVIATIONS | 7 |
| 3. RESPONSIBLE PARTIES | 9 |
| 4. AMENDMENTS AND UPDATES | 10 |
| 5. MILESTONES | 12 |
| 6. RATIONALE AND BACKGROUND | 13 |
| 7. RESEARCH QUESTION AND OBJECTIVES | 14 |
| 8. RESEARCH METHODS | 14 |
| 8.1. Study design | 14 |
| 8.2. Setting. | 14 |
| 8.2.1. Inclusion criteria | 14 |
| 8.2.1.1. COLUMBUS trial | 15 |
| 8.2.1.2. Flatiron Health data | 15 |
| 8.2.2. Exclusion criteria | 16 |
| 8.3. Variables | 17 |
| Table 1. Key exposures, outcomes, and patient baseline characteristics | 17 |
| 8.4. Data sources | 19 |
| 8.5. Study size | 20 |
| 8.6. Data management | 20 |
| 8.7. Data analysis | 21 |
| 8.7.1. Analysis of baseline characteristics | 21 |
| 8.7.2. Unadjusted comparison of OS between treatment groups | 21 |
| 8.7.3. Imputation of missing data on baseline characteristics | 21 |
| 8.7.4. Adjusted comparison of OS between treatment groups | 22 |
| 8.7.5. Exploratory analyses of PFS | 22 |
| 8.8. Quality control | 23 |
| 8.9. Strengths and limitations of the research methods | 23 |
| 8.10. Other aspects | 24 |
| O DEOTECTION OF UTIMAN SUBJECTS | 25 |



| 9.1. Patient information | 25 |
|---|---|
| 9.2. Patient consent. | 25 |
| 9.3. Institutional review board (IRB)/Independent ethics committee (IEC) | 25 |
| 9.4. Ethical conduct of the study | 25 |
| 10. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | 26 |
| 11. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | 27 |
| 12. REFERENCES | 28 |
| 13. LIST OF TABLES | 29 |
| 14. LIST OF FIGURES | 29 |
| ANNEX 1. LIST OF STAND-ALONE DOCUMENTS | 29 |
| ANNEX 2. ADDITIONAL INFORMATION | 29 |
| APPENDIX: TABLE SHELLS | 30 |
| Appendix Table 1: Baseline patient characteristics, by treatment group | 30 |
| Appendix Table 2: Kaplan-Meier analyses comparing OS between treatment group | s .32 |
| Appendix Table 3: Unadjusted and adjusted hazard ratios comparing OS between treatment groups | 32 |



## 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| 1L | First-line |
| AE | Adverse event |
| AJCC | American Joint Committee on Cancer |
| BMI | Body mass index |
| BRAF | v-Raf murine sarcoma viral oncogene homolog B protein |
| CI | Confidence interval |
| CTD | Clinical trial data |
| DAB+TRAM | Dabrafenib + Trametinib |
| ECOG | European Cooperative Oncology Group |
| EHR | Electronic health record |
| ENCO+BINI | Encorafenib + Binimetinib |
| FDA | Food and Drug Administration |
| GPP | Good Pharmacoepidemiology Practices |
| GRACE | Good Research for Comparative Effectiveness |
| HIPAA | Health Insurance Portability and Accountability Act |
| HR | Hazard ratio |
| ICD-9 | International Classification of Diseases 9th Revision |
| ICD-10 | International Classification of Diseases 10th Revision |
| IEC | Independent Ethics Committee |
| Ю | Immunotherapy |
| IRB | Institutional Review Board |
| ISPE | International Society for Pharmacoepidemiology |
| ISPOR | International Society for Pharmacoeconomics and Outcomes Research |
| KM | Kaplan-Meier |
| LDH | Lactate dehydrogenase |
| LOT | Line of therapy |



| MEK | Mitogen-activated protein kinase (MAPK) kinase |
|----------|------------------------------------------------|
| MICE | Multiple imputation by chained equations |
| NDI | National Death Index |
| NI | Non-interventional |
| OS | Overall survival |
| PFS | Progression free survival |
| RECIST | Response Evaluation Criteria in Solid Tumours |
| RWD | Real-world data |
| SMR | Society of Melanoma Research |
| TT | Targeted therapy |
| US | United States |
| VEM+COBI | Vemurafenib + Cobimetinib |



## 3. RESPONSIBLE PARTIES

# Principal Investigator(s) of the Protocol

| Name, degree(s) | Job Title | Affiliation | Address |
|---|---|---|---|
| Kristina Chen, PharmD | Director, Braftovi/<br>Mektovi (Melanoma) | Pfizer, Inc. | 1 Portland Street,<br>Cambridge, MA, 02139 |
| Gautam Sajeev, ScD | Vice President | Analysis Group, Inc. | 111 Huntington Avenue,<br>14th Floor, Boston, MA<br>02199 |
| James Signorovitch,<br>PhD | Managing Principal | Analysis Group, Inc. | 111 Huntington Avenue,<br>14 <sup>th</sup> Floor, Boston, MA<br>02199 |



#### 4. AMENDMENTS AND UPDATES

Significant updates have been made to the data source and analytical approach compared to the original OCEANMIST protocol submission. Below, we provide a high-level overview of the key differences with additional details described in Sections 5-8 and Section 12 below.

# Data Source Updates

• In this study, data for encorafenib plus binimetinib patients will be pooled from the phase 3 COLUMBUS trial and the Flatiron Health real-world database to maximize sample size. In contrast, the original study design, only used encorafenib plus binimetinib data from Flatiron Health. This pooling is justified based on the empirical consistency in OS outcomes across COLUMBUS and Flatiron Health after harmonizing key patient selection criteria, adjusting for differences in baseline characteristics, and imputing missing data on baseline characteristics (HR = 1.03, 95% CI: 0.53, 1.54; p=0.90), described in study C4221035.

## Analytical Approach Updates

- To ensure identification of patient populations in Flatiron that are comparable to patients in the COLUMBUS trial, key patient selection criteria related to age, ECOG performance score, history of brain metastasis and prior use of immunotherapy and targeted therapies from the COLUMBUS trial will be applied to all treatment groups in Flatiron Health.
- To ensure that representation of each targeted therapy from the real-world data was as comprehensive as possible and that patients were followed from treatment initiation consistent with the COLUMBUS trial, patients included in each treatment cohort will be required to have index dates (i.e., treatment initiation dates) that were on or after the dates of FDA approval of that targeted therapy in metastatic melanoma (specifically, 09 January 2014 for DAB+TRAM, 10 November 2015 for VEM+COBI and 27 June 2018 for ENCO+BINI). This is in contrast to the original approach, which defined the follow-up period for all cohorts as beginning from 20 November 2015. This could have led to the exclusion of some patients initiating DAB+TRAM before approval, and could potentially inadvertently include off-label usage of ENCO+BINI.
- For the real-world cohorts, patient baseline characteristics will be obtained from visits ≤3 months prior to the index date, with data from visits closest in time to the index date being used as available. In contrast, in the original protocol, to maximize availability of baseline characteristics, the 'baseline' period was allowed to include visits up to 6 months prior to treatment initiation. The decision to use a stricter definition of baseline here was based on clinical input that certain baseline characteristics of interest (e.g., ECOG PS) are best assessed closest to the index date, despite potential for increased missingness. To address missingness, imputation of baseline characteristics was conducted as described below.



- Key clinical characteristics like ECOG and LDH were missing at baseline for 40-60% of
  patients in the original study cohort, which would have hampered ability to adjust for
  potential confounding due to these factors. To address missingness, we will impute data
  using multiple imputation by chained equations prior to conducting adjusted analyses.
  Imputation models will be based on baseline characteristics that would be considered in
  adjusted models for OS.
- Inverse probability of treatment weighting without any imputation was proposed in the
  original study design to account for baseline differences. Instead, we will use
  multivariable Cox proportional hazards models fit to each of the imputed dataset and
  combined results across all imputations. This approach is preferred as it allows us to
  assess how included covariates are associated with OS in our final models, in addition to
  estimating differences between the treatments of interest.
- Comparisons of OS and PFS were stratified by first-line and second-line of therapy in the
  original study design. Analyses conducted in this revised protocol will not be stratified by
  line of therapy to allow for a larger sample size to compare OS and PFS across targeted
  therapy treatment cohorts. A line of therapy variable will be included in Cox proportional
  hazard models, which can facilitate future analyses of comparative effectiveness by line
  of therapy if required.



# 5. MILESTONES

| Milestone | Planned date |
|---|---|
| Amendment to study protocol | 19 May 2023 |
| Completion of statistical analyses | 7 June 2023 |
| Abstract submission to Society for Melanoma Research (SMR) 2023 Congress | 21 June 2023 |
| Final study report | 21 July 2023 |



#### 6. RATIONALE AND BACKGROUND

Melanoma, caused when malignant cancer cells form in melanocytes, is the fifth most common cancer in the United States (US) and the deadliest form of skin cancer. Incidence of melanoma has been increasing over recent decades, with the overall incidence rate of 229.1 cases per million person based on recent estimates. Based on American Cancer Society estimates, there were an estimated 99,780 new cases of melanoma and ~7,650 deaths from melanoma in the US in 2022. 1-3

Approximately 9% of melanoma patients are diagnosed with regional spread to lymph nodes and 4% are diagnosed with metastatic disease. Compared to patients with localized melanoma, patients with metastatic melanoma have poorer prognosis and worse outcomes, which can be further worsened by the presence of v-Raf murine sarcoma viral oncogene homolog B protein (BRAF) mutations. The BRAF protein plays an important role in normal cell growth, proliferation, differentiation, and survival. The presence of BRAF V600 mutations, found in ~40–60% of melanoma cases, can lead to sustained mitogen-activated protein kinase (MAPK) kinase (MEK) pathway signaling, resulting in tumor growth and progression.

Recommended treatment options for metastatic melanoma include immunotherapy (IO), which attempts to stimulate host responses to effectuate tumor destruction, and targeted therapies (TT), which inhibit molecular pathways to prevent tumor growth and maintenance. The discovery of targeted therapy as a treatment for melanoma has emerged as a milestone development in oncological research. In 2018, the US Food and Drug Administration (FDA) approved the use of encorafenib (BRAFTOVI®) in combination with binimetinib (MEKTOVI®) for the treatment of patients with unresectable or metastatic melanoma with a BRAF V600E or V600K mutation (as detected by an FDA-approved test) based on the pivotal phase 3 COLUMBUS trial. This accompanied existing BRAF-/MEK-inhibitor therapies including dabrafenib plus trametinib (FDA approval 10 November 2015).

There is increasing interest in evaluating comparative effectiveness of BRAF-/MEK-inhibitor therapies. In a recent study, we showed that overall survival (OS) for metastatic BRAFV600-mutant melanoma patients was similar across the COLUMBUS trial and real-world practice data from the Flatiron Health database (Hazard Ratio [HR] = 0.94, 95% Confidence Interval [CI]: 0.43, 1.45) after harmonizing key patient selection criteria, adjusting for differences in baseline characteristics, and imputing missing data on baseline characteristics. Given this empirical consistency in OS outcomes, pooling patients across these settings can be justified and allows for a larger sample size for assessment of comparative effectiveness of encorafenib + binimetinib versus other targeted therapies. To that end, this study will expand on this prior work and compare OS between patients receiving encorafenib + binimetinib in the pooled Phase 3 COLUMBUS trial and the Flatiron Health Electronic Health Records (EHR) database versus patients receiving other targeted therapies. Baseline profiles of patients will also be compared to characterize differences in patients receiving different therapies and adjustments will be made for



differences across treatment groups in baseline factors associated with OS. Missingness for key baseline characteristics will be addressed using a validated multiple imputation approach.<sup>12</sup>

# 7. RESEARCH QUESTION AND OBJECTIVES

### Primary Objective

To compare OS between patients with metastatic BRAFV600-mutant melanoma initiating encorafenib plus binimetinib (ENCO+BINI) versus dabrafenib plus trametinib (DAB+TRAM) or vemurafenib plus cobimetinib (VEM+COBI)

# Exploratory Objective

To compare progression free survival (PFS) between patients with metastatic BRAFV600mutant melanoma initiating ENCO+BINI versus DAB+TRAM or VEM+COBI

This objective is designated as exploratory as, unlike for OS, differences in assessment of PFS between clinical trial data (CTD) and real-world data (RWD) settings may exist that preclude valid comparisons of this outcome across these settings. Suitability of comparative analyses of PFS will be determined following additional exploration to characterize number and frequency of assessments of PFS, and further analyses of comparability of PFS outcomes across trial and real-world settings.

#### 8. RESEARCH METHODS

#### 8.1. Study design

This is a retrospective cohort study comparing OS outcomes between patients with BRAFV600-mutant metastatic melanoma initiating ENCO+BINI versus DAB+TRAM or VEM+COBI. Comparisons will be adjusted for differences in baseline characteristics across treatment groups, and account for missing data on adjustment factors. PFS will also be investigated as an exploratory endpoint, subject to comparability of PFS outcome assessment between clinical trial and real-world settings.

#### 8.2. Setting

Patients with BRAFV600-mutant metastatic melanoma initiating treatment with ENCO+BINI, DAB+TRAM or VEM+COBI.

#### 8.2.1. Inclusion criteria

Inclusion criteria that will be used to identify patients initiating the targeted therapies of interest are provided separately for the clinical trial and real-world data sources below.



#### 8.2.1.1. COLUMBUS trial

Key inclusion criteria in the COLUMBUS trial were:

- Histologically confirmed diagnosis of locally advanced, unresectable, or metastatic cutaneous melanoma or unknown primary melanoma
- American Joint Committee on Cancer (AJCC) disease stage of IIIB, IIIC, IVM1a, IVM1b, or IVM1c at trial enrolment
- Presence of BRAF V600E or V600K mutation in tumor tissue prior to enrollment
- At least 18 years of age at randomization
- Eastern Cooperative Oncology Group (ECOG) status of 0 or 1 at randomization
- Treatment naive or had progressed on or after previous first-line (1L) immunotherapy at randomization with no prior BRAF- or MEK-inhibitor therapy in the adjuvant setting

Patients from the COLUMBUS trial included in this analysis will be those patients:

Randomized to ENCO+BINI arm of the trial to receive 450mg once daily encorafenib
and 45mg twice daily binimetinib combination therapy

#### 8.2.1.2. Flatiron Health data

Pfizer has contracted with Flatiron for a custom data extract containing information on patients with advanced melanoma. Eligibility criteria applied to the Flatiron custom data received by Pfizer include:

- Diagnosed with melanoma based on International Classification of Disease 9th and 10<sup>th</sup> Revisions (ICD-9: 172.x; ICD-10: C43x, D03x) and ≥2 visits on different days in the Flatiron database on or after January 1, 2011.
- Clinically confirmed diagnosis of melanoma with pathologic stages III or IV at initial diagnosis or earlier stage disease with a first locoregional or distant recurrence on or after January 1, 2011.
- Age ≥18 years at the time of advanced melanoma diagnosis.
- Evidence of ≥1 BRAF positive test result at any time based on laboratory or genetic analysis results.
- Treatment with ≥1 BRAF-inhibitor (i.e., encorafenib, dabrafenib, vemurafenib) and treatment with ≥1 MEK-inhibitor (i.e., binimetinib, trametinib, cobimetinib) in 1L or 2L line of therapy (LOT), as defined per Flatiron's LOT business rules.



 Earliest LOT containing a BRAF- and MEK-inhibitor ≥3 months prior to data cutoff (defined as 30 September 2021)

Key inclusion criteria from the COLUMBUS trial will be applied to the Flatiron RWD population to align the populations to the extent possible between the CTD and RWD sources. The sample of patients from the Flatiron Health EHR data for this study will be identified using the following additional criteria applied to the custom data cut received from Flatiron:

- At least 18 years of age at the index date
- Confirmed BRAF V600E or V600K activating mutation reported in the data based on laboratory or genetic analysis results
- Treatment-naive or had previous 1L IO at index date in the therapeutic setting, based on review of medication orders or administration prior to the index date.
- ECOG status of 0 or 1 at the index date

The following criteria will be additionally used to identify patients receiving each of the treatments of interest:

- ENCO+BINI treatment group: At least 1 order or administration of ENCO+BINI treatment after the diagnosis of metastatic melanoma and after 27 June 2018 (FDA approval date for ENCO+BINI for use in patients with metastatic melanoma).
- DAB+TRAM treatment group: At least 1 order or administration of DAB+TRAM treatment after the diagnosis of metastatic melanoma and after 09 January 2014 (FDA approval date for DAB+TRAM for use in patients with metastatic melanoma).
- VEM+COBI treatment group: At least 1 order or administration of VEM+COBI treatment after the diagnosis of metastatic melanoma and after 10 November 2015 (FDA approval date for VEM+COBI for use in patients with metastatic melanoma).

The index date in each treatment group will be the date of treatment initiation.

#### 8.2.2. Exclusion criteria

Patients meeting any of the following criteria will not be included in the study:

- Patients with prior BRAF- or MEK-inhibitor therapy
- Patients with ECOG performance status ≥ 2 (at the time of randomization for patients from COLUMBUS, during the baseline period for patients in Flatiron EHR)
- Patients with a history of leptomeningeal metastases including brain, spinal cord, or nervous system metastases (based on brain MRI or CT scan with contrast-enhanced brain MRI as the preferred assessment in COLUMBUS and based on the following



diagnostic codes in Flatiron EHR: ICD-9-CM: 198.3, 198.4 or ICD-10-CM: C79.31, C79.32, C79.40, C79.49) prior to index

For RWD patients, concurrent enrollment in a clinical trial.

#### 8.3. Variables

Table 1 provides a summary of exposure, outcome, and patient baseline characteristics that will be evaluated within the study.

Table 1. Key exposures, outcomes, and patient baseline characteristics

| Variable | Role | Data source(s) | Operational definition/categories |
|---|---|---|---|
| Treatment group<br>(ENCO+BINI,<br>DAB+TRAM,<br>VEM+COBI) | Exposure | COLUMBUS<br>trial data;<br>Flatiron EHR | Indicates whether patients initiated ENCO+BINI,<br>DAB+TRAM or VEM+COBI treatment |
| os | Primary Outcome | COLUMBUS<br>trial data, | In the COLUMBUS trial data, defined as the time from the date of randomization to the date of death due to any cause; if death is not observed, patients will be censored at the date of last contact or the data analysis cut-off date (e.g., 15 September 2020), whichever occurs first |
| | 7 Timary Sutcome | Flatiron | In Flatiron EHR, will be defined as the time from the index<br>date to the date of death; patients without a date of death<br>will be censored at their last known activity date (e.g., the<br>last clinical note date) or the end of the follow-up period,<br>whichever occurs first |
| | PFS Exploratory Outcome | COLUMBUS<br>trial data,<br>Flatiron her | In the COLUMBUS trial data, defined as the time from the date of randomization to the date of the first documented disease progression or death due to any cause, whichever occurred first; if a patient did not have an event at the analysis cut-off date, PFS will be censored at the date of the last adequate tumour assessment |
| PFS | | | In Flatiron EHR, will be defined as the time from the index date to either the date of first disease progression event or death in the absence of progression; patients without disease progression or death will be censored at the last date the patient could have been assessed for progression (e.g., the last clinical note date) or the data analysis cut-off date (e.g., 30 September 2021), whichever occurs first |
| Age at baseline<br>(years) | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data<br>Flatiron EHR | Patient age; defined at the time of study randomization for<br>COLUMBUS trial data and at the time of treatment<br>initiation for Flatiron EHR |
| Sex | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | Male, Female, Intersex, or Unknown/Missing |



| Race | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | Asian, Black, White, Other/Multi-Race, or<br>Unknown/Missing |
|---|---|---|---|
| Body mass index<br>(BMI) at index | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | Defined as weight (in kg) divided by squared height (in m²) |
| ECOG at index | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | 0, 1, Unknown/Missing; defined during the baseline period<br>of both the COLUMBUS trial data and Flatiron EHR |
| BRAF mutation<br>status | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | V600E, V600K, Unknown/Missing |
| AJCC disease stage<br>at initial melanoma<br>diagnosis | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | 0, I, II, III, IV, or Unknown/Missing; defined at initial<br>melanoma diagnosis for COLUMBUS trial data and<br>Flatiron EHR |
| AJCC disease stage<br>at treatment<br>initiation | Baseline Characteristic | COLUMBUS<br>trial data | IIIB, IIIC, IVM1a, IVM1b, or IVM1c; defined at treatment initiation in the COLUMBUS trial data. Not available in the Flatiron EHR |
| Lactate<br>dehydrogenase<br>(LDH) at index | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | Evaluated in units per liter (U/L) and defined at trial<br>baseline in COLUMBUS trial and during the baseline<br>period in Flatiron EHR |
| Time from initial<br>melanoma diagnosis<br>to metastatic disease | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | Duration (in months) from melanoma diagnosis to the<br>development of metastatic disease |
| Time from<br>metastatic<br>melanoma diagnosis<br>to treatment<br>initiation | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | Duration (in months) from metastatic melanoma diagnosis<br>to the initiation of treatment |
| Year of treatment initiation | Baseline Characteristic | COLUMBUS<br>trial data;<br>Flatiron EHR | Calendar year when treatment was initiated |
| Region | Baseline Characteristic | COLUMBUS<br>trial data;<br>Flatiron EHR | Europe, North America, Australia, Other, or Missing |
| Treatment<br>experience in the<br>therapeutic setting | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | Indicates whether patients received targeted therapy as<br>first-line treatment (e.g., Treatment naïve) or as second-<br>line treatment after a prior line of immunotherapy<br>treatment (e.g., Prior 1L IO therapy) |
| Prior systemic<br>therapies in the<br>adjuvant setting | Baseline Characteristic<br>/Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | Indicates whether patients previously received systemic therapy (e.g., prior surgery, radiotherapy, immunotherapy, or chemotherapy) before initiating treatment |
| Prior surgery in the adjuvant setting | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | Indicates whether patients previously used surgery to reduce/remove tumors as a form of treatment |
| Prior radiotherapy<br>in the adjuvant<br>setting | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | Indicates whether patients underwent radiotherapy among those receiving prior systemic therapy |



| Prior IO or<br>chemotherapy in the<br>adjuvant setting | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | Indicates whether patients underwent chemotherapy or immunotherapy among those receiving prior systemic therapy |
|---|---|---|---|
| Number of LOTs<br>after TT treatment<br>initiation | Baseline Characteristic /<br>Potential Confounder | COLUMBUS<br>trial data;<br>Flatiron EHR | Indicates the number of LOTs occurring after treatment initiation $(0, 1, \ge 2$ , or Missing) |
| Number of organs<br>involved | Baseline Characteristic | COLUMBUS<br>trial data;<br>Flatiron EHR | Indicates number of organs involved or sites of metastases at baseline (1, 2, or ≥3), with all patients having at least 1 site given diagnosis of metastatic disease. This data was collected and reported in COLUMBUS. In Flatiron EHR, it will be derived based on counting the number of distinct sites recorded as having metastases based on ICD codes. |
| Presence of lung<br>metastases | Baseline Characteristic | COLUMBUS<br>trial data;<br>Flatiron EHR | Indicates whether patients had lung metastases. This data was collected and reported in COLUMBUS. In Flatiron EHR, it will be derived based on having ICD codes reflecting presence of lung or respiratory organ metastases (ICD-9: 197, 197.1; ICD-10: C78.01, C78.02, C78.1, C78.2, C78.30, C78.39). |
| Presence of liver<br>metastases | Baseline Characteristic | COLUMBUS<br>trial data;<br>Flatiron EHR | Indicates whether patients had liver metastases. This data was collected and reported in COLUMBUS. In Flatiron EHR, it will be derived based on having ICD codes reflecting presence of liver metastases (ICD-9: 197.7; ICD-10: C78.7) |
| Presence of other<br>metastases | Baseline Characteristic | COLUMBUS<br>trial data;<br>Flatiron EHR | Indicates whether patients had presence of other metastases (e.g., adrenal glands, bone, digestive tract/system, kidney, lymph nodes, reproductive organs, or unspecified sites). This data was collected and reported in COLUMBUS. In Flatiron EHR, it will be derived based on having ICD codes reflecting presence of other metastases (ICD-9: 196, 196.1, 196.2, 196.3, 196.5, 196.6, 196.8, 196.9, 197.4, 197.5, 197.6, 197.8, 198, 198.5, 198.7, 198.89; ICD-10: C77.0, C77.1, C77.2, C77.3, C77.4, C77.5, C77.8, C77.9, C78.4, C78.5, C78.6, C78.80, C78.89, C79.00, C79.01, C79.02, C79.11, C79.51, C79.52, C79.60, C79.61, C79.62, C79.70, C79.71, C79.72, C79.81, C79.89, C79.9) |

#### 8.4. Data sources

## COLUMBUS trial

COLUMBUS was a two-part, multicenter, randomized, open-label, Phase 3 clinical trial. <sup>10</sup> Part 1 of the trial investigated the effectiveness and safety of three treatment regimens in patients with locally advanced unresectable or metastatic BRAFV600-mutant metastatic melanoma who were treatment naïve or whose cancer had progressed after 1L IO. In Part 1 of the trial, patients were randomized to one of three treatment arms: 1) 450mg once daily encorafenib and 45mg twice daily binimetinib (n=192), 2) 960mg twice daily vemurafenib (n=191) and 3) 300mg once daily



encorafenib (n=194). Randomization was stratified by AJCC disease stage (IIIB, IIIC, IVM1a, IVM1b, or IVM1c), ECOG performance status (0, 1), and BRAFV600 mutation profile (V600E, V600K). Progression-free survival was the primary endpoint in the trial, while OS was one of the secondary endpoints. Patients were enrolled in Part 1 of the trial between 30 December 2013 through 10 April 2015.

The ENCO+BINI arm of Part 1 of the trial will be used in this study (database lock date: 15 September 2020). Part 2 of the trial compared encorafenib 300mg once daily plus binimetinib 45mg twice daily versus encorafenib 300mg once daily alone and will not be considered.

#### Flatiron Health EHR

The Flatiron Health EHR database is a longitudinal, de-identified real-world database derived from EHRs collected in US cancer clinics. The database covers more than 2.6 million active cancer patients treated at over 800 sites of care across 4 US census regions. Patient-level data includes both structured (diagnosis, demographics, laboratory values, biomarker information, drug orders, visits, etc.) and unstructured (physician notes, radiology, and pathology reports, etc.) sources. Data on death is drawn from structured or unstructured data fields in the EHR, and publicly available sources of mortality including the US Social Security Death Index, and commercial obituary data. <sup>13</sup>

Pfizer has contracted with Flatiron for a custom data extract containing information on patients with advanced melanoma who received treatment with BRAF- or MEK-inhibitor therapies. Patients meeting the eligibility criteria defined for this study will be obtained from this custom data extract as described in Section 8.2 and used in all analyses.

#### 8.5. Study size

The number of patients eligible for the study will be determined in accordance with the sample selection conducted per the criteria described in Section 8.2.

#### 8.6. Data management

Clean, patient-level datasets for COLUMBUS and Flatiron Health data will be generated for use throughout the study. This process will entail basic exploratory checks to ensure data integrity, cleaning and reformatting the raw data as needed, and creating variables for all key study measures. All data will be stored and maintained on a secure encrypted non-cloud-based server and accessed over a secure internal private wide area network. The data will be made accessible only to individuals working on the current study. No attempt will be made to identify individual patients, hospitals, or physicians. Analyses will be conducted using SAS version 9.4 and/or R version 4.1.0 or later.



#### 8.7. Data analysis

## 8.7.1. Analysis of baseline characteristics

Patient baseline characteristics at or prior to the index visit will be summarized for all treatment groups. Patient characteristics to be summarized will be based on availability in both data sources and clinical input. A list of characteristics expected to be summarized is provided in Table 1.

Baseline characteristics will be summarized at the index date if measured at that time. In the Flatiron data, for baseline characteristics that are not measured at the index date, the closest available measure to the index date within a baseline period will be used. Informed by clinical input and considerations of data availability, the baseline period will be defined as a 3-month time window prior to and including the index date.

Patient baseline characteristics will be summarized descriptively using mean (with standard deviation) and median (with interquartile range) for continuous variables and count (with proportions) for categorical variables. Missingness for each baseline characteristic (at the index date or within the baseline period) will also be summarized.

# 8.7.2. Unadjusted comparison of OS between treatment groups

OS will be defined as described in Section 8.3. OS will be summarized for each treatment group (i.e., ENCO+BINI [pooled across COLUMBUS and Flatiron EHR], DAB+TRAM and VEM+COBI). An unadjusted comparison of OS across treatment groups will be conducted using Kaplan-Meier (KM) analyses. OS over time in these treatment groups will be plotted and compared using a log-rank test, with median survival time and survival proportions reported at selected time points (e.g., 6 months, 1 year, 2 years). Hazard ratios for OS comparing ENCO+BINI relative to DAB+TRAM and VEM+COBI will be estimated based on a univariable Cox proportion hazards model. The proportional hazards assumption will be assessed using tests of Schoenfeld residuals. 14

## 8.7.3. Imputation of missing data on baseline characteristics

Previous analyses of the Flatiron data have found that there are moderate to large amounts of missing data on baseline characteristics such as ECOG performance score and LDH. <sup>12</sup> As analyses restricted to patients with non-missing data are highly likely to be biased, imputation of missing data on key baseline characteristics is needed to ensure that adjusted analyses of OS between the trial and RWD settings are based on all eligible patients.

In this study, multiple imputation by chained equations (MICE)<sup>15</sup> will be used to impute missing data on baseline characteristics. Briefly, the MICE method imputes data for a missing patient characteristic based on iterative regressions of observed data for that characteristic on observed and imputed values of other baseline characteristics. This process will be repeated for each



characteristic until stable estimates are obtained, and the entire procedure will be repeated so that multiple datasets with imputed values for baseline characteristics are created.

Baseline characteristics to be imputed will include ECOG performance score, LDH, and other clinical or demographic characteristics (e.g., race, BMI, etc.). Additional variables (e.g., age, sex, AJCC diagnosis, time from MM diagnosis to treatment initiation, time from initial diagnosis of melanoma to metastatic disease, number of organs at baseline, metastatic sites, treatments in the therapeutic setting, treatments in the adjuvant setting) will be considered for inclusion in the MICE procedure based on their relevance for adjustment and degree of missingness in the study sample. As recommended in the literature, the MICE approach will be used to create multiple datasets (e.g., 100 datasets) with imputed values, which will be used and combined in subsequent analyses. <sup>15</sup>

Missing data on baseline characteristics will be imputed for all treatment groups. Analyses of baseline characteristics described in Section 8.7.1 will be repeated for each imputed dataset, and then summarized across all imputed datasets.

#### 8.7.4. Adjusted comparison of OS between treatment groups

Finally, an adjusted comparison of OS across treatment groups (i.e., ENCO+BINI [pooled across COLUMBUS and Flatiron EHR], DAB+TRAM and VEM+COBI) will be conducted. Hazard ratios will be estimated based on a multivariable Cox proportional hazard model, adjusting for key baseline characteristics known or expected to be related to OS in metastatic melanoma (e.g., age, sex, race, BMI, ECOG, LDH, time from initial melanoma diagnosis to metastatic disease, time from metastatic diagnosis to treatment initiation, treatment experience in the therapeutic setting, prior IO/chemotherapy in the adjuvant setting, prior surgery in the adjuvant setting). Specific adjustment factors listed here may be revised based on expert clinical input.

The adjusted analyses will be conducted in each of the datasets with imputed baseline characteristic values in turn. Log-hazard ratios for OS comparing treatment with ENCO+BINI relative to DAB+TRAM and VEM+COBI each imputed dataset will be obtained, and summary HRs obtained by pooling results across all imputed datasets will be generated using Rubin's rules. <sup>16</sup>

## 8.7.5. Exploratory analyses of PFS

Analyses assessing PFS will also be explored. PFS will be defined as described in Section 8.3. PFS will be summarized for all treatment groups.

Suitability of comparative analyses of PFS between treatment groups will be determined following additional data exploration to characterize number and frequency of assessments of PFS available in these settings, and discussion of comparability of the assessment of disease progression in RWD vs CTD. If analyses of PFS are deemed suitable based on these evaluations,



unadjusted and adjusted comparisons of PFS will be conducted using the methods described in Sections 8.7.2 and 8.7.4.

#### 8.8. Quality control

Best practice guidelines will be followed to ensure project quality, including structured organization of project materials (e.g., data extracts, statistical software programs, output tables) and standard internal audit process. The audit process both confirms the validity of the analytical approach and ensures that all programs and results are accurate.

# 8.9. Strengths and limitations of the research methods

The strengths of this study include:

- Key inclusion criteria with respect to diagnosis, disease stage, age, BRAFV600 mutation and ECOG status in the COLUMBUS trial will be applied to the Flatiron RWD to the extent possible to obtain a comparable group of patients across both settings
- Adjustment will be made for multiple baseline characteristics to mitigate bias due to potential differences in these characteristics across the treatment groups
- Concerns about differences in outcome assessment across trial and RWD settings are
  mitigated for OS given the availability of a real-world mortality endpoint in the Flatiron
  RWD that has high sensitivity, specificity, positive predictive values, negative predictive
  values and agreement when compared against the National Death Index (NDI), the goldstandard source for mortality data in the US.<sup>17</sup>

The limitations of this study include the following:

- Application of the COLUMBUS trial inclusion criterion requiring at least 1 measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria will not be implemented due to absence in Flatiron EHR of systematic radiographic imaging to assess tumor response as required by RECIST.
- While adjustment will be made for available baseline characteristics across treatment
  groups, differences due to factors that were not adjusted for may still contribute to
  observed differences in OS between settings. For instance, data on number and sites of
  metastases, while systematically collected in the COLUMBUS trial, can only be derived
  based on ICD codes in Flatiron EHR. Based on clinical input, data on number and sites
  of metastases will very likely be underestimated in the Flatiron EHR, and not
  comparable to the corresponding data from COLUMBUS, precluding adjustment for
  these variables.



- The analysis conducted here is analogous to an 'intent-to-treat' perspective, and therefore will not account for potential differences in adherence and post-baseline treatments between trial and real-world settings.
- The COLUMBUS trial was a multi-national trial that recruited patients from 160+ sites in 28 countries, and therefore covers a broader range of geographies than the US-based Flatiron RWD; differences in background care across geographies and care settings may contribute to differences in outcomes between the CTD and RWD.

## 8.10. Other aspects

Not applicable.



#### 9. PROTECTION OF HUMAN SUBJECTS

#### 9.1. Patient information

This study involves data that exist in anonymized structured format and contain no patient personal information.

#### 9.2. Patient consent

As this study involves anonymized structured data, which according to applicable legal requirements do not contain data subject to privacy laws, obtaining informed consent from patients by Pfizer is not required.

## 9.3. Institutional review board (IRB)/Independent ethics committee (IEC)

This retrospective database analysis does not involve the collection, use, or transmittal of individually identifiable data. As such, the study falls within the definition of exempt research under 45 CFR 46.104(d)(4)(ii) and IRB approval is not required. Because the dataset does not include individually identifiable health information under 45 CFR 164.514, Health Insurance Portability and Accountability Act (HIPAA) requirements do not apply.

## 9.4. Ethical conduct of the study

The study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value and rigor and follow generally accepted research practices described in in Guidelines for Good Pharmacoepidemiology Practices (GPP) issued by the International Society for Pharmacoepidemiology (ISPE), Good Practices for Outcomes Research issued by the International Society for Pharmacoeconomics and Outcomes Research (ISPOR), and the Good Research for Comparative Effectiveness (GRACE) Principles. 18-20



# 10. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

This study involves electronic health records data that exist as structured data by the time of study start or a combination of existing structured data and unstructured data, which will be converted to structured form during the implementation of the protocol solely by a computer using automated/algorithmic methods, such as natural language processing.

In these data sources, individual patient data are not retrieved or validated, and it is not possible to link (i.e., identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (i.e., identifiable patient, identifiable reporter, a suspect product, and event) cannot be met.



#### 11. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

In the event of any prohibition or restriction imposed (e.g., clinical hold) by an applicable competent authority in any area of the world, or if the investigator, Analysis Group, is aware of any new information which might influence the evaluation of the benefits and risks of a Pfizer product, Pfizer should be informed immediately.

Based on the analysis results and discussions with Pfizer, an abstract and/or manuscript may be prepared. If feasible, an abstract will be submitted to the Society for Melanoma Research (SMR) 2023 conference. A study report summarizing the background, objectives, methods, results, and conclusion of the study will be prepared.



#### 12. REFERENCES

- SEER Cancer Stat Facts: Melanoma of the Skin. National Cancer Institute. https://seer.cancer.gov/statfacts/html/melan.html
- ACS. American Cancer Society. Cancer Facts & Figures 2021. 2021.
- Society AC. Cancer Facts & Figures 2022. American Cancer Society.
- Paulson KG, Gupta D, Kim TS, et al. Age-Specific Incidence of Melanoma in the United States. JAMA Dermatology. 2020;156(1):57. doi:10.1001/jamadermatol.2019.3353
- Holderfield M, Deuker MM, McCormick F, McMahon M. Targeting RAF kinases for cancer therapy: BRAF-mutated melanoma and beyond. *Nature Reviews Cancer*. 2014;14(7):455-467. doi:10.1038/nrc3760
- 6. Ny L, Hernberg M, Nyakas M, et al. BRAF mutational status as a prognostic marker for survival in malignant melanoma: a systematic review and meta-analysis. *Acta Oncologica*. 2020;59(7):833-844. doi:10.1080/0284186x.2020.1747636
- Vanneman M, Dranoff G. Combining immunotherapy and targeted therapies in cancer treatment. *Nature reviews cancer*. 2012;12(4):237-251.
- 8. Bhatia P, Friedlander P, Zakaria EA, Kandil E. Impact of BRAF mutation status in the prognosis of cutaneous melanoma: an area of ongoing research. *Annals of translational medicine*. 2015;3(2)
- FDA approves encorafenib and binimetinib in combination for unresectable or metastatic melanoma with BRAF mutations. 2018. https://www.fda.gov/drugs/resources-informationapproved-drugs/fda-approves-encorafenib-and-binimetinib-combination-unresectable-ormetastatic-melanoma-braf
- Dummer R, Ascierto PA, Gogas HJ, et al. Encorafenib plus binimetinib versus vemurafenib or encorafenib in patients with BRAF-mutant melanoma (COLUMBUS): a multicentre, open-label, randomised phase 3 trial. *The Lancet Oncology*. 2018;19(5):603-615.
- 11. Pocock SJ. The combination of randomized and historical controls in clinical trials. Journal of chronic diseases. 1976;29(3):175-188.
- Signorovitch J, Moshyk A, Zhao J, et al. Overall survival in the real-world and clinical trials: a case study validating external controls in advanced melanoma. *Future Oncol*. Apr 2022;18(11):1321-1331. doi:10.2217/fon-2021-1054
- Curtis MD, Griffith SD, Tucker M, et al. Development and Validation of a High-Quality Composite Real-World Mortality Endpoint. *Health Serv Res*. Dec 2018;53(6):4460-4476. doi:10.1111/1475-6773.12872
- Grambsch PM, Therneau TM. Proportional hazards tests and diagnostics based on weighted residuals. *Biometrika*. 1994;81(3):515-526.
- 15. White IR, Royston P, Wood AM. Multiple imputation using chained equations: Issues and guidance for practice. *Stat Med.* Feb 20 2011;30(4):377-99. doi:10.1002/sim.4067
- Rubin DB. Multiple imputation for nonresponse in surveys. vol 81. John Wiley & Sons;
   2004.
- Zhang Q, Gossai A, Monroe S, Nussbaum NC, Parrinello CM. Validation analysis of a composite real-world mortality endpoint for patients with cancer in the United States. *Health* Serv Res. Dec 2021;56(6):1281-1287. doi:10.1111/1475-6773.13669



- 18. Berger ML, Sox H, Willke RJ, et al. Good practices for real-world data studies of treatment and/or comparative effectiveness: recommendations from the joint ISPOR-ISPE Special Task Force on real-world evidence in health care decision making. *Value in Health*. 2017;20(8):1003-1008.
- International Society for Pharmacoeconomics and Outcomes Research I. ISPOR Good Practices Reports. Accessed 28 March 2023, https://www.ispor.org/heor-resources/goodpractices
- Public Policy Committee ISoP. Guidelines for good pharmacoepidemiology practice (GPP). Pharmacoepidemiology and drug safety. 2016;25(1):2-10.

#### 13. LIST OF TABLES

| Table | Description |
|---|---|
| Table 1. Key exposures, outcomes, and patient | Table summarizing exposure, outcome, and |
| baseline characteristics in the treatment groups | patient baseline characteristics that will be |
| | evaluated within the study. |
| Table 2. Kaplan-Meier analyses comparing OS | Table summarizing KM analyses from the |
| between treatment groups | ENCO+BINI, DAB+TRAM and VEM+COBI |
| | treatment groups |
| Table 3. Unadjusted and adjusted hazard ratios | Table summarizing hazard ratios comparing |
| comparing OS between treatment groups | ENCO+BINI to the DAB+TRAM and |
| | VEM+COBI treatment groups |

#### 14. LIST OF FIGURES

None.

#### ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

None.

## ANNEX 2. ADDITIONAL INFORMATION

Not applicable.



## APPENDIX: TABLE SHELLS

# Appendix Table 1: Baseline patient characteristics, by treatment group

| | ENCO+BINI | VEM+COBI | DAB+TRAM |
|---|---|---|---|
| | N = | N = | N = |
| Demographic Characteristics | | | |
| Age at baseline (years) | | | |
| Mean (SD) | | | |
| Median (IQR) | | | |
| Sex, n (%) | | | |
| Female | | | |
| Male | | | |
| Missing, n (%) | | | |
| Race, n (%) | | | |
| White/Caucasian | | | |
| Black/African American | | | |
| Asian | | | |
| Native American or Pacific Islander | | | |
| Other | | | |
| Missing | | | |
| BMI (kg/m²) | | | |
| Mean (SD) | | | |
| Median (IQR) | | | |
| Missing, n (%) | | | |
| Year of treatment initiation, n (%) | | | |
| 2014 | | | |
| 2015 | | | |
| 2016 | | | |
| 2017 | | | |
| 2018 | | | |
| 2019 | | | |
| 2020 | | | |
| 2021 | | | |
| Region, n (%) | | | |
| North America | | | |
| Europe | | | |
| Australia | | | |
| Other | | | |
| Missing | | | |
| Disease-Related Characteristics | | | |
| Number of organs involved (metastatic sites | s) at baseline, n (%) | | |
| 1 | | | |
| 2 | | | |
| ≥3 | | | |
| Missing | | | |
| Lung metastasis, n (%) | | | |
| No | | | |
| Yes | | | |



| Missing | | |
|---|---|---|
| Liver metastasis, n (%) | | |
| No | | |
| Yes | | |
| Missing | | |
| Other metastasis, n (%) | | |
| No | | |
| Yes | | |
| Missing | | |
| Time from initial melanoma diagnosis to | metastatic disease (months | ) |
| Mean (SD) | | |
| Median (IQR) | | |
| Missing, n (%) | | |
| Time from metastatic melanoma diagnos | is to treatment initiation (m | onths) |
| Mean (SD) | | |
| Median (IQR) | | |
| Missing, n (%) | | |
| BRAF mutation status, n (%) | | |
| V600E | | |
| V600K | | |
| ECOG performance status, n (%) | | |
| 0 | | |
| 1 | | |
| ≥2 | | |
| Missing | | |
| AJCC stage at initial melanoma diagnosis, | n (%) | |
| 0 | | |
| I | | |
| П | | |
| III | | |
| IV | | |
| Unknown | | |
| Missing | | |
| AJCC stage at treatment initiation, n (%) | | |
| Stage IIIC | | |
| Stage IV | | |
| Missing | | |
| LDH categories, n (%) | | |
| ≤ULN | | |
| > ULN | | |
| Missing | | |
| Treatment-Related Characteristics | | |
| Treatment experience in the therapeutic setting, n (%) | | |
| Treatment naive | | |
| Prior 1L IO therapy | | |
| Prior systemic therapies in the adjuvant setting, n (%) | | |
| Yes | | |



| N- | T |
|---|---|
| No | |
| Prior IO or chemotherapy in the adjuvan | Prior IO or chemotherapy in the adjuvant setting, n (%) |
| Yes | |
| No | |
| Prior surgery in the adjuvant setting, n ( | Prior surgery in the adjuvant setting, n (%) |
| Yes | |
| No | |
| Number of LOTs after targeted therapy, n (%) | |
| 0 | |
| 1 | |
| ≥2 | |
| Missing | |

# Appendix Table 2: Kaplan-Meier analyses comparing OS between treatment groups

| | ENCO+BINI | VEM+COBI | DAB+TRAM |
|---|---|---|---|
| | N = | N = | N = |
| Summary of deaths, censoring | | | |
| and median survival | | | |
| Death, n (%) | | | |
| Censored, n (%) | | | |
| Median follow-up (95% CI) | | | |
| Median OS (95% CI) | | | |
| Kaplan-Meier based estimates of % | of patients remaining | | |
| alive at different time points | | | |
| 6 Months | | | |
| 12 Months | | | |
| 18 Months | | | |
| 24 Months | | | |
| 30 Months | | | |
| 36 Months | | | |

Appendix Table 3: Unadjusted and adjusted hazard ratios comparing OS between treatment groups

Results from adjusted models in Appendix Table 3 will be based on multiple imputation via multivariate imputation by chained equations. Expected adjustment factors are listed below; specific functional forms/categorization of adjustment factors will be based on the data.

| | Unadjusted model | Adjusted model |
|------------------------|------------------|----------------|
| | HR (95% CI) | HR (95% CI) |
| Treatment group | | |
| DAB+TRAM vs. ENCO+BINI | | |
| (ref) | | |



| VEM+COBI vs. ENCO+BINI |
|---------------------------------|
| (ref) |
| Adjustment factors |
| Age (years) |
| Male vs female |
| Asian race vs. White |
| Other race vs. White |
| Unknown race vs. White |
| BMI (kg/m²) |
| ECOG (1 vs. 0) |
| LDH (>ULN vs. ≤ULN) |
| Treatment naïve vs. prior 1L |
| IO treatment |
| Prior IO/chemotherapy (Yes |
| vs. No) |
| Prior surgery (Yes vs. No) |
| Time from initial melanoma |
| diagnosis to metastatic disease |
| Time from metastatic disease |
| to treatment initiation |